CLINICAL TRIAL: NCT02581865
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of NBI-98854 in Adult Subjects With Tourette Syndrome
Brief Title: Safety and Efficacy Study of NBI-98854 in Adults With Tourette Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-98854-1505
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Results first posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — valbenazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placebo (Placebo Comparator): Placebo administered once daily for 8 weeks
  Interventions: Drug: Placebo
- Dose Group 1 (Experimental): Fixed dose administered once daily for 8 weeks
  Interventions: Drug: NBI-98854
- Dose Group 2 (Experimental): Fixed dose administered once daily for 8 weeks
  Interventions: Drug: NBI-98854

INTERVENTIONS:
Drug: NBI-98854
  Arms: Dose Group 1; Dose Group 2
Drug: Placebo
  Arms: Placebo

SUMMARY:
Phase 2, double-blind, placebo-controlled study to assess the safety and efficacy of NBI-98854 administered once daily (qd) for a total of 8 weeks of treatment. This study will enroll approximately 90 male and female subjects clinically diagnosed with Tourette Syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Have a clinical diagnosis of Tourette Syndrome (TS)
2. Have at least moderate tic severity
3. Have TS symptoms that impair school, occupational, and/or social function
4. If using maintenance medication(s) for TS or TS spectrum diagnoses (e.g. obsessive-compulsive disorder [OCD], Attention-Deficit Hyperactivity Disorder [ADHD]), be on stable doses
5. Be in good general health
6. Have a negative urine drug screen for amphetamines, barbiturates, benzodiazepine, phencyclidine, cocaine, or opiates, and a negative alcohol screen
7. Subjects of childbearing potential who do not practice total abstinence must agree to use hormonal or two forms of nonhormonal contraception (dual contraception) consistently during the screening, treatment and follow-up periods of the study

Exclusion Criteria:

1. Have an active, clinically significant unstable medical condition within 1 month prior to screening
2. Have a known history of long QT syndrome or cardiac tachy-arrhythmia
3. Have a known history of neuroleptic malignant syndrome
4. Have a cancer diagnosis within 3 years prior to screening (some exceptions allowed)
5. Have an allergy, hypersensitivity, or intolerance to VMAT2 inhibitors
6. Have a known history of substance dependence, substance (drug) or alcohol abuse
7. Have a significant risk of suicidal or violent behavior
8. Are currently pregnant or breastfeeding
9. Have initiated Comprehensive Behavioral Intervention for Tics (CBIT) during the screening period or at baseline or plan to initiate CBIT during the study
10. Have received an investigational drug within 30 days before screening or plan to use an investigational drug (other than NBI-98854) during the study
11. Have a blood loss ≥550 mL or donated blood within 30 days prior to screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (30):
  - Long Beach, California
  - National City, California
  - San Bernardino, California
  - San Diego, California
  - Upland, California
  - Gainesville, Florida
  - Hialeah, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Boston, Massachusetts
  - Natick, Massachusetts
  - St Louis, Missouri
  - Nashua, New Hampshire
  - Summit, New Jersey
  - Albany, New York
  - Manhasset, New York
  - New York, New York
  - Staten Island, New York
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Norristown, Pennsylvania
  - Nashville, Tennessee
  - Dallas, Texas
  - Irving, Texas
  - Orem, Utah
  - Salt Lake City, Utah
  - Kirkland, Washington
  - Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled participants (male and female) with a diagnosis of Tourette Syndrome through Diagnostic and Statistical Manual of Mental Disorders, 4th or 5th Editions (DSM-IV or -V) from approximately 40 study centers in the United States
Groups:
- NBI-98854 40 mg: Fixed dose of NBI-98854 40 mg administered once daily for 8 weeks
- NBI-98854 80 mg: NBI-98854 80 mg dose will be titrated in a blinded fashion (subjects will receive 40 mg for the first week followed by 80 mg for the remainder of the 8-week treatment period)
Period: Overall Study
Arm/Group | Placebo | NBI-98854 40 mg | NBI-98854 80 mg
Started | 40 | 42 | 42
Completed | 36 | 35 | 26
Not Completed | 4 | 7 | 16

BASELINE CHARACTERISTICS:
Population: the intent-to-treat (ITT) analysis set, that includes all randomized subjects who received at least one dose of study drug, have postbaseline safety data & have at least one post randomization Yale Global Tic Severity Scale (YGTSS) Total Tic Score (TTS) value at a scheduled visit or mapped early termination (ET) visit during 8-week treatment period
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | NBI-98854 40 mg | NBI-98854 80 mg | Total
Number analyzed (Participants) | 39 | 41 | 40 | 120
Age, Continuous [Mean (Full Range); unit: years] | 37.2 [18 to 62] | 34.1 [18 to 64] | 34.1 [18 to 61] | 35.1 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 15 | 40
  Male | 23 | 32 | 25 | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 4 | 9
  Not Hispanic or Latino | 36 | 39 | 36 | 111
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race: Asian | 1 | 0 | 1 | 2
  Race: Black or African American | 2 | 2 | 1 | 5
  Race: White | 34 | 39 | 34 | 107
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Race: Other | 0 | 0 | 0 | 0
  Race: American Indian or Alaska Native, White | 2 | 0 | 1 | 3
  Race: Black or African American, White | 0 | 0 | 1 | 1
  Race: White, Other: German | 0 | 0 | 1 | 1
  Race: Other: Thai/White | 0 | 0 | 1 | 1
Body mass index (BMI) at Screening [Mean (Full Range); unit: kg/m^2 (kilogram/meter^2)] | 28.69 [18.8 to 40.0] | 28.75 [19.2 to 38.3] | 29.01 [18.2 to 43.5] | 28.82 [18.2 to 43.5]
Yale Global Tic Severity Scale (YGTSS) Total Tic Score (TTS) [Mean (Full Range); unit: Score on scale] — The YGTSS is designed to rate the overall severity of motor and phonic tic symptoms across a range of dimensions: number, frequency, intensity, complexity, and interference. The YGTSS was administered by the investigator (or qualified designee) using a computer-based structured clinical interview. The TTS is the sum of the 5 motor tic items and the 5 phonic (vocal) tic items and ranges from 0 to 50, with higher scores representing greater severity
  Score on scale | 32.1 [16 to 47] | 31.6 [17 to 45] | 30.0 [19 to 45] | 31.2 [16 to 47]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in the YGTSS TTS
Description: The YGTSS is designed to rate the overall severity of motor and phonic tic symptoms across a range of dimensions: number, frequency, intensity, complexity, and interference. The YGTSS was administered by the investigator (or qualified designee) using a computer-based structured clinical interview. The TTS is the sum of the 5 motor tic items and the 5 phonic (vocal) tic items and ranges from 0 to 50, with higher scores representing greater severity
Time Frame: Baseline, Week 8
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Least Squares Mean (Standard Error)
Groups:
- NBI-98854 80 mg: NBI-98854 80 mg dose titrated in a blinded fashion (subjects will receive 40 mg for the first week followed by 80 mg for the remainder of the 8-week treatment period)
Arm/Group | Placebo | NBI-98854 40 mg | NBI-98854 80 mg
Number analyzed (Participants) | 37 | 35 | 27
Least Squares Mean (Standard Error) | -6.1 (1.1) | -7.4 (1.7) | -8.0 (1.1)
Statistical Analysis 1: Comparison: Placebo vs NBI-98854 40 mg; Test type: Superiority; p = 0.4326, Mixed Models Analysis; Mean Difference (Net) = -1.4, 95% CI 2-sided [-4.9 to 2.1], Standard Error of Mean 1.8
Statistical Analysis 2: Comparison: Placebo vs NBI-98854 80 mg; Test type: Superiority; p = 0.1835, Mixed Models Analysis; Mean Difference (Net) = -2.5, 95% CI 2-sided [-6.2 to 1.2], Standard Error of Mean 1.9

2. Secondary Outcome: Clinical Global Impression of Change Tourette Syndrome (CGI-TS)-Improvement Score at Week 8
Description: The CGI-TS-Improvement scale is used to assess overall improvement since the initiation of study drug dosing on a 7-point scale. Each of the CGI-TS-Improvement response categories was assigned a numerical score as follows: 1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = Not changed; 5 = Minimally worse; 6 = Much worse; 7 = Very much worse.
Time Frame: Week 8
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | NBI-98854 40 mg | NBI-98854 80 mg
Number analyzed (Participants) | 37 | 36 | 27
score on a scale | 3.2 (0.2) | 3.0 (0.2) | 2.6 (0.1)
Statistical Analysis 1: Comparison: Placebo vs NBI-98854 40 mg; Test type: Superiority; p = 0.3812, ANOVA; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.7 to 0.3], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Placebo vs NBI-98854 80 mg; Test type: Superiority; p = 0.0146, ANOVA; Mean Difference (Net) = -0.7, 95% CI 2-sided [-1.2 to -0.1], Standard Error of Mean 0.3

3. Secondary Outcome: Change From Baseline to Week 8 in the Clinical Global Impression of Tics (CGI-Tics)-Severity Score
Description: The CGI-Tics-Severity scale is used to assess overall severity on a 7-point scale. Each of the CGI-Tics-Severity response categories was assigned a numerical score as follows: 1 = Normal, not at all ill; 2 = Borderline ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; 7 = Among the most extremely ill patient.
Time Frame: Baseline, Week 8
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- NBI-98854 80 mg: NBI-98854 80 mg dose titrated in a blinded fashion (subjects received 40 mg for the first week followed by 80 mg for the remainder of the 8-week treatment period)
Arm/Group | Placebo | NBI-98854 40 mg | NBI-98854 80 mg
Number analyzed (Participants) | 37 | 36 | 27
score on a scale | -0.8 (0.2) | -1.0 (0.2) | -1.0 (0.1)
Statistical Analysis 1: Comparison: Placebo vs NBI-98854 40 mg; Test type: Superiority; p = 0.3065, Mixed Models Analysis; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.6 to 0.2], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Placebo vs NBI-98854 80 mg; Test type: Superiority; p = 0.2052, Mixed Models Analysis; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.7 to 0.2], Standard Error of Mean 0.2

4. Secondary Outcome: Change From Baseline to Last Visit in the Rush Video-based Tic Rating Scale (RTRS) Total Score
Description: A modified RTRS was used in this study that includes short video recordings to measure 5 tic variables: number of body areas affected, frequency of motor and phonic tics, and severity of motor and phonic tics. The RTRS total score is calculated as the sum of the 5 domain scores, and ranges from 0 to 20, with higher scores representing greater severity. The final on-treatment visit was used in subjects who discontinued prior to Week 8.
Time Frame: Baseline, Week 8
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | NBI-98854 40 mg | NBI-98854 80 mg
Number analyzed (Participants) | 39 | 41 | 40
score on a scale | -1.9 (0.7) | -3.0 (0.6) | -3.6 (0.6)
Statistical Analysis 1: Comparison: Placebo vs NBI-98854 40 mg; Test type: Superiority; p = 0.2215, ANCOVA; Mean Difference (Net) = -1.0, 95% CI 2-sided [-2.7 to 0.6], Standard Error of Mean 0.8
Statistical Analysis 2: Comparison: Placebo vs NBI-98854 80 mg; Test type: Superiority; p = 0.0566, ANCOVA; Mean Difference (Net) = -1.6, 95% CI 2-sided [-3.3 to 0.0], Standard Error of Mean 0.9

5. Secondary Outcome: Change From Baseline to Week 8 in the YGTSS Global Tic Severity Score
Description: The YGTSS Global Tic Severity score is the sum of the YGTSS TTS and the YGTSS Impairment score and ranges from 0 to 100, with higher scores representing greater severity.
Time Frame: Baseline, Week 8
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- NBI-98854 80 mg: NBI-98854 80 mg dose titrated in a blinded fashion (subjects will receive 40 mg for the first week followed by 80 mg for the remainder of the 8-week treatment period
Arm/Group | Placebo | NBI-98854 40 mg | NBI-98854 80 mg
Number analyzed (Participants) | 37 | 35 | 27
score on a scale | -15.0 (2.6) | -16.2 (3.5) | -19.1 (2.9)
Statistical Analysis 1: Comparison: Placebo vs NBI-98854 40 mg; Test type: Superiority; p = 0.5689, Mixed Models Analysis; Mean Difference (Net) = -2.2, 95% CI 2-sided [-9.8 to 5.4], Standard Error of Mean 3.8
Statistical Analysis 2: Comparison: Placebo vs NBI-98854 80 mg; Test type: Superiority; p = 0.2320, Mixed Models Analysis; Mean Difference (Net) = -4.8, 95% CI 2-sided [-12.8 to 3.1], Standard Error of Mean 4.0

6. Secondary Outcome: Change From Baseline to Week 8 in the Premonitory Urge for Tics Scale (PUTS) Total Score
Description: The PUTS is an instrument for quantifying the premonitory urge phenomena associated with tics. It consists of 9 items, each of which is scored on a 4-point scale (1=not at all true, 2=a little true, 3=pretty much true, 4=very much true). The PUTS total score is calculated as the sum of the scores for the 9 items. The maximum possible total score is 36.
Time Frame: Baseline, Week 8
Population: The analysis population include intent-to-treat (ITT):all subjects in the safety analysis set with at least one post-randomization TTS value reported at a scheduled visit or mapped Early Termination (ET) visit during the treatment period.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- NBI-98854 80 mg: NBI-98854 80 mg dose titrated in a blinded fashion (subjects will received 40 mg for the first week followed by 80 mg for the remainder of the 8-week treatment period).
Arm/Group | Placebo | NBI-98854 40 mg | NBI-98854 80 mg
Number analyzed (Participants) | 37 | 36 | 27
score on a scale | -1.2 (0.7) | -0.8 (0.9) | -0.6 (0.9)
Statistical Analysis 1: Comparison: Placebo vs NBI-98854 40 mg; Test type: Superiority; p = 0.4515, Mixed Models Analysis; Mean Difference (Net) = -0.8, 95% CI 2-sided [-3.0 to 1.3], Standard Error of Mean 1.1
Statistical Analysis 2: Comparison: Placebo vs NBI-98854 80 mg; Test type: Superiority; p = 0.6289, Mixed Models Analysis; Mean Difference (Net) = -0.5, 95% CI 2-sided [-2.8 to 1.7], Standard Error of Mean 1.1

ADVERSE EVENTS:
Time Frame: Up to 10 Weeks
Description: All TEAEs,whether observed by investigator,reported by subject,noted from lab. findings,or identified by other means, were recorded from time subject signed ICF until subject's follow-up visit(Week 10 or ET).
  The analysis set include all subjects who are randomized to a treatment group and dispensed study drug, with two exclusions:(a)subjects who withdraw from study & return all previously dispensed study drug with all doses present,&(b) subjects who have no postbaseline safety data collected.
Groups:
- NBI-98854 80 mg: NBI-98854 80 mg dose was titrated in a blinded fashion (subjects will receive 40 mg for the first week followed by 80 mg for the remainder of the 8-week treatment period
Arm/Group | Placebo | NBI-98854 40 mg | NBI-98854 80 mg
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/42 | 2/42
Other Adverse Events (participants affected / at risk) | 8/40 | 22/42 | 32/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | NBI-98854 40 mg (N=42) | NBI-98854 80 mg (N=42)
Septic shock (Infections and infestations) | 0 | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=40) | NBI-98854 40 mg (N=42) | NBI-98854 80 mg (N=42)
Somnolence (Nervous system disorders) | 1 | 8 | 9
Akathisia (Nervous system disorders) | 0 | 1 | 10
Headache (Nervous system disorders) | 2 | 6 | 2
Lethargy (Nervous system disorders) | 0 | 2 | 3
Sedation (Nervous system disorders) | 1 | 1 | 4
Disturbance in attention (Nervous system disorders) | 0 | 0 | 3
Fatigue (General disorders) | 1 | 5 | 7 — The Organ system term used to generate the source table is General disorders and administration site conditions
Anxiety (Psychiatric disorders) | 1 | 1 | 4
Insomnia (Psychiatric disorders) | 0 | 0 | 5
Nausea (Gastrointestinal disorders) | 1 | 1 | 4
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI has the right to publish results provided such publication does not violate confidentiality or IP provisions within the contract with the Sponsor. Prior to submission for publication or presentation of results, the PI must provide the Sponsor time for review. The Sponsor can request the PI to withhold or remove information from all publications. For a multi-center study, any publication of results by the PI shall not be made before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-06-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT02581865/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT02581865/SAP_001.pdf